CLINICAL TRIAL: NCT02067494
Title: Myofascial Release and Kinesiotaping on Disability, Pain, Automic Nervous System and Oxidative Stress Indicators in Chronic Low Back Pain: A Randomized Controlled Clinical Trial
Brief Title: Myofascial Release and Kinesio Taping on Autonomic Nervous System in Low Back Pain
Acronym: I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, Lecturer, Universidad de Almeria
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UAL-032
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Low Back Pain; Chronic Disease
Keywords: Low Back Pain; Chronic Pain; Manual Therapy; Randomized Clinical Trial; Bandages
MeSH Terms: conditions — Low Back Pain; Chronic Disease; Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Myofascial Soft Tissue Release (Experimental): * Protocol: Myofascial release on thoracolumbar fascia, Myofascial release on diaphragm, Myofascial release in the psoas fascia, Indirect Myofascial release restrictions in the public area, Myofascial release in lumbo-sacral decompression, Myofascial release on sacrum, and Myofascial release on the lumbar fascia.
  * Myofascial release assisted the paravertebral fascia.
  Interventions: Other: Myofascial Soft Tissue Release
- Kinesio taping treatment (Active Comparator): Two bands in "I", with anchor onset in sacrum, on paravertebral muscles. Furthermore a strip will be applies on correction space point of maximum pain.
  Interventions: Other: Kinesio taping treatment

INTERVENTIONS:
Other: Myofascial Soft Tissue Release — Protocol: Myofascial release on thoracolumbar fascia, Myofascial release on diaphragm, Myofascial release in the psoas fascia, Indirect Myofascial release restrictions in the public area, Myofascial release in lumbo-sacral decompression, Myofascial release on sacrum, and Myofascial release on the lumbar fascia.
  Arms: Myofascial Soft Tissue Release
Other: Kinesio taping treatment — Two bands in "I", with anchor onset in sacrum, on paravertebral muscles. Furthermore a strip will be applies on correction space point of maximum pain.
  Arms: Kinesio taping treatment

SUMMARY:
The purpose of this current randomized clinical trial is to determine the effects of myofascial soft tissue release and kinesio taping on disability, pain, quality of life, autonomic nervous system and oxidative stress indicators in chronic low back pain.

DETAILED DESCRIPTION:
Design: Randomized Clinical Trial. Objective: to determine the effects of myofascial soft tissue release and kinesio taping on pain, disability, quality of life, and autonomic nervous system indicators.

Methods and Measures: sixty-four individuals will be randomly assigned to one of two groups.

Intervention: For 10-week, the group 1 will undergo treatment comprising a myofascial soft tissue release protocol (1/week) and the group 2 will recieve a kinesio taping treatment (1/week).

Main Outcome Measures: Intensity of pain, disability, quality of life, biochemical stimation intertitial fluid, body mass indicators, hormonal indicators, indicators of autonomic nevous system, and indicators of oxidative stress will be collected in both groups at baseline, 10 weeks and 15 weeks after the last intervention. Baseline demographic and clinical variables will be examined between both groups with an independent Student t-test for continuous data. Separate 2x3 model ANOVA with time (baseline, 10 weeks and 15 weeks) as the within-subjects factor, group will be to determine the effects of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Score ≥ 4 on the Roland Morris Disability Questionnaire.
* Low Back Pain for ≥ 3 months.
* Not undergoing another physical therapy treatment.

Exclusion Criteria:

* Disease of the central or peripheral nervous system.
* Having previously undergone manual therapy.
* Contraindication to low back manual therapy.
* A history of spinal surgery.
* Treatment with corticosteroid in the past two weeks.
* Clinical sign of radiculopathy
* Presence of Stenosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Roland Morris Disability Questionnaire (RMDQ) | At baseline, 10 weeks and 15 weeks
  This is a self-reported questionnaire consisting of 24 items reflecting limitations in different activities of daily living attributed to low back pain including walking, bending over, sitting, lying down, dressing, sleeping, self-care and daily activities

SECONDARY OUTCOMES:
Change form baseline in Visual Analogue Scale | At baseline, 10 weeks and 15 weeks
  A 10-point Numerical Pain Scale (0: no pain, 10: maximum pain) assesses the intensity of pain.
Change from baseline in Lifestyle Indicators | At baseline, 10 weeks and 15 weeks
  Estimation of interstitial fluid biochemistry and measure the following indicators: body mass, hormonal, autonomic nervous system and oxidative stress.
Change from baseline on Neural Network Analysis | At baseline, 10 weeks and 15 weeks
  Analysis of the projection on the spine and segmental innervation projection.
Change from baseline on Quality of Life | At baseline, 10 weeks and 15 weeks
  SF-36 Health questionnaire scores range from 0 to 100% and indicate the self-perceived health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Adelaida Castro-Sánchez, Lecturer, Principal Investigator — Universidad de Almeria
Locations (1):
- Universidad de Almeria, Almería, Almería, Spain

REFERENCES:
- [Background] Nijs J, Meeus M, Cagnie B, Roussel NA, Dolphens M, Van Oosterwijck J, Danneels L. A modern neuroscience approach to chronic spinal pain: combining pain neuroscience education with cognition-targeted motor control training. Phys Ther. 2014 May;94(5):730-8. doi: 10.2522/ptj.20130258. Epub 2014 Jan 30. PMID 24481595
- [Background] Taylor JB, Goode AP, George SZ, Cook CE. Incidence and risk factors for first-time incident low back pain: a systematic review and meta-analysis. Spine J. 2014 Oct 1;14(10):2299-319. doi: 10.1016/j.spinee.2014.01.026. Epub 2014 Jan 23. PMID 24462537
- [Background] Adorno ML, Brasil-Neto JP. Assessment of the quality of life through the SF-36 questionnaire in patients with chronic nonspecific low back pain. Acta Ortop Bras. 2013 Jul;21(4):202-7. doi: 10.1590/S1413-78522013000400004. PMID 24453669
- [Background] Biely SA, Silfies SP, Smith SS, Hicks GE. Clinical observation of standing trunk movements: what do the aberrant movement patterns tell us? J Orthop Sports Phys Ther. 2014 Apr;44(4):262-72. doi: 10.2519/jospt.2014.4988. Epub 2014 Jan 22. PMID 24450372
- [Background] Kramer CD, Koch WH, Fritz JM. Development and outcomes of a program to translate the evidence for spinal manipulation into physical therapy practice. J Man Manip Ther. 2013 Nov;21(4):177-86. doi: 10.1179/2042618613Y.0000000036. PMID 24421630
- [Background] Bae SH, Lee JH, Oh KA, Kim KY. The effects of kinesio taping on potential in chronic low back pain patients anticipatory postural control and cerebral cortex. J Phys Ther Sci. 2013 Nov;25(11):1367-71. doi: 10.1589/jpts.25.1367. Epub 2013 Dec 11. PMID 24396190
- [Background] Alvarez-Alvarez S, Jose FG, Rodriguez-Fernandez AL, Gueita-Rodriguez J, Waller BJ. Effects of Kinesio(R) Tape in low back muscle fatigue: randomized, controlled, doubled-blinded clinical trial on healthy subjects. J Back Musculoskelet Rehabil. 2014;27(2):203-12. doi: 10.3233/BMR-130437. PMID 24284272
- [Background] Added MA, Costa LO, Fukuda TY, de Freitas DG, Salomao EC, Monteiro RL, Costa Lda C. Efficacy of adding the Kinesio Taping method to guideline-endorsed conventional physiotherapy in patients with chronic nonspecific low back pain: a randomised controlled trial. BMC Musculoskelet Disord. 2013 Oct 24;14:301. doi: 10.1186/1471-2474-14-301. PMID 24156687
- [Background] Castro-Sanchez AM, Lara-Palomo IC, Mataran-Penarrocha GA, Fernandez-Sanchez M, Sanchez-Labraca N, Arroyo-Morales M. Kinesio Taping reduces disability and pain slightly in chronic non-specific low back pain: a randomised trial. J Physiother. 2012;58(2):89-95. doi: 10.1016/S1836-9553(12)70088-7. PMID 22613238
- [Background] Lee JH, Yoo WG. Application of posterior pelvic tilt taping for the treatment of chronic low back pain with sacroiliac joint dysfunction and increased sacral horizontal angle. Phys Ther Sport. 2012 Nov;13(4):279-85. doi: 10.1016/j.ptsp.2011.10.003. Epub 2011 Dec 8. PMID 23068906